CLINICAL TRIAL: NCT06121648
Title: Effect of Hydrotherapy on the Balance and Fatigue of Multiple Sclerosis Patients
Brief Title: Effect of Hydrotherapy on Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantinos Chandolias, Post Doc Researcher, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6006
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Hydrotherapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: 2 groups
  1. water group
  2. land group
Who Masked: Participant
Masking Description: closed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water Group (Experimental): Static and dynamic balance, breathing, combined breathing and movement activities.
  Interventions: Other: hydrotherapy
- Land Group (Active Comparator): Intervention program focused on balance and gait.
  Interventions: Other: neurological physiotherapy

INTERVENTIONS:
Other: hydrotherapy — 30 degrees temperature pool balance and breathing therapy
  Arms: Water Group
Other: neurological physiotherapy — Balance and neurological physiotherapy on land
  Arms: Land Group

SUMMARY:
The purpose of this work was to investigate the effect of a hydrotherapy program on the balance and fatigue of patients with multiple sclerosis. it is a fact that hydrotherapy has an effect on the rehabilitation and treatment of people with balance problems.

DETAILED DESCRIPTION:
26 patients with multiple sclerosis participated in the present research, who were divided into 2 intervention groups, one in the sea and one on land. The intervention program had a duration of 2 months with a frequency of 2 times a week for both groups. The interventions were performed by specialized therapists. All participants were assessed before and after the intervention using the BBS and MFIS scales.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with RR-type (relapsing-remitting) multiple sclerosis by MS ( multiple sclerosis) expert neurologists, and Expanded Disability Status Scale (EDSS) cit 10 Score of 1-3.7 participated in this study.

Exclusion Criteria:

* older than 45 years; EDSS Score>3,7; primary progressive MS; acute or chronic physical or psychological disorders; participation in less than 12 of the 16 hydrotherapy sessions; common contraindications for hydrotherapy as cardiovascular disease, allergy etc.,

Ages: 23 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
BBS scale | 2 months
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
MFIS scale | 2 months
  The total MFIS score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamía, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.Beck CA, Metz LM, Svenson LW, Patten SB. Regional variation of multiple sclerosis prevalence in Canada. Mult Scler 2005;11(5):516-9. 2.Corvillo I, Varela E, Armijo F, Alvarez-Badillo A, Armijo O, Maraver F. Efficacy of aquatic therapy for multiple sclerosis: a systematic review. Eur J Phys Rehabil Med 2017 [ahead of print]. 3.Multiple sclerosis: Hope through research. https://www.ninds.nih.gov/ Disorders/Patient-Caregiver-Education/Hope-Through-Research/MultipleSclerosis-Hope-Through-Research. Accessed October 1, 2018. 4. Ms prevalence: National multiple sclerosis society. https://www.nationalmssociety.org/About-the-Society/MS-Prevalence. Accessed October 2, 2018, 2018. 10 Kurtzke JF. Rating neurologic impairment in multiple sclerosis. Neurology 1983;33:1444. Alikhajeh, Y., Hosseini, S. R. A., & Moghaddam, A. (2012). Effects of hydrotherapy in static and dynamic balance among elderly men. Procedia-Social and Behavioral Sciences, 46, 2220-2224. Bekiari, M., Iakovidis, P., Lytras, D., Chatziprodromidou, I. P., & Dimitros, E. (2021). The effect of hydrotherapy on the symptoms and functional characteristics of multiple sclerosis patients. Int J Phys Educ Sport Heal, 8(2), 191-197. Castro-Sánchez, A. M., Matarán-Peñarrocha, G. A., Lara-Palomo, I., Saavedra-Hernández, M., Arroyo-Morales, M., & Moreno-Lorenzo, C. (2012). Hydrotherapy for the treatment of pain in people with multiple sclerosis: a randomized controlled trial. Evidence-based complementary and alternative medicine, 2012. Dixon, J., Hatton, A. L., Robinson, J., Gamesby-Iyayi, H., Hodgson, D., Rome, K., ... & Martin, D. J. (2014). Effect of textured insoles on balance and gait in people with multiple sclerosis: an exploratory trial. Physiotherapy, 100(2), 142-149. Genova, H., Dacosta-Aguayo, R., Goverover, Y., Smith, A., Bober, C., & DeLuca, J. (2020). Effects of a Single Bout of Aquatic Exercise on Mood in Multiple SclerosisA Pilot Study. International Journal of MS Care, 22(4), 173-177. Hammill, H. V., Ellapen, T. J., Strydom, G. L., & Swanepoel, M. (2018). The benefits of hydrotherapy to patients with spinal cord injuries. African journal of disability, 7(1), 1-8. Kahraman, T., Rasova, K., Jonsdottir, J., Medina, C. S., Kos, D., Coote, S., ... & Kalron, A. (2022). The impact of the COVID-19 pandemic on physical therapy practice for people with multiple sclerosis: A multicenter survey study of the RIMS network. Multiple Sclerosis and Related Disorders, 62, 103799. Kargarfard, M., Etemadifar, M., Baker, P., Mehrabi, M., & Hayatbakhsh, R. (2012). Effect of aquatic exercise training on fatigue and health-related quality of life in patients with multiple sclerosis. Archives of physical medicine and rehabilitation, 93(10), 1701-1708. Kubsik-Gidlewska, A. M., Klimkiewicz, P., Klimkiewicz, R., Janczewska, K., & Woldańska-Okońska, M. Z. (2017). Rehabilitation in multiple sclerosis. Advances in Clinical and Experimental Medicine, 26(4). Lambeck, J. (2017). Hydrotherapy in adult neurology. EWAC Medical http://www. ewac. com. Accessed, 10. Mooventhan, A., & Nivethitha, L. (2014). Scientific evidence-based effects of hydrotherapy on various systems of the body. North American journal of medical sciences, 6(5), 199. Ormstad, H., Simonsen, C. S., Broch, L., Maes, M., Anderson, G., & Celius, E. G. (2020). Chronic fatigue and depression due to multiple sclerosis: Immune-inflammatory pathways, tryptophan catabolites and the gut-brain axis as possible shared pathways. Multiple sclerosis and related disorders, 46, 102533. Tan, Z., Liu, H., Yan, T., Jin, D., He, X., Zheng, X., ... & Tan, C. (2014). The effectiveness of functional electrical stimulation based on a normal gait pattern on subjects with early stroke: a randomized controlled trial. BioMed research international, 2014.